CLINICAL TRIAL: NCT00693953
Title: Using the Digital EEG Spectral Analysis in Assessing Neuroelectrical Processing Abnormalities in Autism
Status: Withdrawn | Type: Observational
Why Stopped: grant was not approved.
Sponsor: Yellen & Associates, Inc. (Other)
Responsible Party: Dr. Andrew G. Yellen, Yellen & Associates, Inc.
Other Study IDs: PA-06-278
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Autistic Disorder; Autism, Early Infantile; Autism, Infantile; Asperger Syndrome
Keywords: Evoked Potentials; Evoked Potentials, Auditory; Evoked Potentials, Visual; Electroencephalography; Brain Mapping
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Year one
- 2: Year two

SUMMARY:
Individuals with Autism Spectrum Disorder will have abnormal DESA® results. Our objective is to use neuroelectrical measures to determine the degree of processing abnormalities in individuals with Autism. The study will survey processing patterns and will locate and evaluate the degree(s) of abnormalities for further study. The abnormal results of comprehensive neuroelectrical evaluations of individuals with Autism when compared to the normative database will provide objective, verifiable, neurophysiological information with which to form novel approaches to the disorder.

DETAILED DESCRIPTION:
The research method will be: gathering, analyzing and utilizing data.

We will observe research subjects through neuroelectrical instrumentation, then, compare results to retrospective information collected from research subjects and a normative database.

A qualified neurologist thoroughly familiar with electrophysiology will interpret the data, and analyze it to explore the abnormalities.

The hypothesis will be evaluated.

We will, then, utilize the results to find data-based forms of treatment for those with the disorder.

ELIGIBILITY:
Inclusion Criteria:

* The study will include children between the ages of five and eighteen, adults from the age of nineteen to twenty-five, and those with the diagnosis of Autism and Autism Spectrum Disorders.

Exclusion Criteria:

* those with mental retardation
* those with any other neurological disorder
* those that cannot sit in a chair for one hundred and fifty minutes
* those that have been previously diagnosed with a seizure disorder
* those who are blind and/or deaf
* those who are not ambulatory
* those who cannot understand English
* those that are not a resident of Los Angeles County

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes individuals with Autism without exclusion on the basis of sex, gender, race or ethnicity. There will be 100 research subjects, with a ratio of four males to one female, and those being approximately sixty-five children and thirty-five adults.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Yellen, PhD, Principal Investigator — President, Yellen & Associates, Inc.; Thomas Schweller, MD, Study Chair — Neurologist
Locations (1):
- Yellen & Associates, Inc., Northridge, California, United States